CLINICAL TRIAL: NCT02677493
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Parallel Phase III Study to Investigate the Immunogenicity and Safety of 'IL-YANG Quadrivalent Influenza Vaccine Inj.' After Intramuscular Administration in Healthy Adult Subjects
Brief Title: Study to Evaluate the Immunogenicity and Safety of 'IL-YANG Quadrivalent Influenza Vaccine Inj.'
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IY_IFEZ_Q301
Record Dates: First submitted 2016-02-03; First posted 2016-02-09 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2020-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IL-YANG Quadrivalent Influenza Vaccine (Experimental): The QIV is included both B strain (Yamagata, Victoria).
  Interventions: Biological: IL-YANG Quadrivalent Influenza Vaccine
- IL-YANG Flu Vaccine Prefilled Syringe (Active Comparator): This TIV is included the B/Yamagata strain, and it was approved for commercial sale by MFDS.
  Interventions: Biological: IL-YANG Flu Vaccine Prefilled Syringe
- IL-YANG Trivalent Influenza Vaccine (Active Comparator): This TIV is included the B/Victoria strain.
  Interventions: Biological: IL-YANG Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: IL-YANG Quadrivalent Influenza Vaccine — A single 0.5mL dose administrated as an intramuscular injection.
  Arms: IL-YANG Quadrivalent Influenza Vaccine
Biological: IL-YANG Flu Vaccine Prefilled Syringe — A single 0.5mL dose administrated as an intramuscular injection.
  Arms: IL-YANG Flu Vaccine Prefilled Syringe
Biological: IL-YANG Trivalent Influenza Vaccine — A single 0.5mL dose administrated as an intramuscular injection.
  Arms: IL-YANG Trivalent Influenza Vaccine

SUMMARY:
This study evaluates the immunogenicity and safety of 'IL-YANG Quadrivalent Influenza Vaccine Inj.' in healthy male and female adults at the age of 19 or older.

DETAILED DESCRIPTION:
In this study, only eligible subjects for the study based on the inclusion/exclusion criteria will be randomized to the following stratification groups by age to receive one dose of the test vaccine, comparator 1, or comparator 2.

* Group A: healthy adults at the age of ≥ 19 and < 65.
* Group B: healthy adults at the age of ≥ 65.

During the study participation, the investigator will assess immunogenicity and safety in subjects. The investigator will perform immunogenicity tests at Visits 1 and 3 (end of study visit) for immunogenicity evaluation (prior to the investigational product vaccination) and instruct subjects to record AEs occurring after the investigational product vaccination for safety assessment.

A blood sample will be collected from a subject who is assigned a subject number. Following an intramuscular injection of 0.5mL investigational product in the deltoid muscle of the shoulder, the subject will have a study visit on Week 4 for blood sampling for antibody titer testing. In addition, a telephone visit will be performed to assess serious AEs (SAEs) up to Day 180 after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women at the age of 19 or older.
* Women of childbearing potential must have a negative pregnancy test (urine HCG) at the screening visit.
* Subjects who were given, and fully understood, the information about the study, and have provided voluntary written informed consent to participate in the study and to comply with all applicable study requirements.

Exclusion Criteria:

* Subjects with known allergy to eggs, chicken, or any components of the study vaccine.
* Subjects who had received an influenza vaccine within the last 6 months prior to study entry.
* Subjects who have immune function disorders including immunodeficiency diseases or relevant family history.
* Subjects who donated blood within 1 week prior to vaccination or plan to donate blood during the period from Day 1 to Month 7 of vaccination.
* Subjects with a history of Guillain-Barre syndrome.
* Subjects with Down's syndrome or cytogenetic disorders.
* Subjects who are considered by the investigator to have difficulties in study participation due to severe chronic diseases (e.g., cardiovascular diseases except controlled hypertension and respiratory diseases with respiratory failure, metabolic diseases, renal function disorders, hemoglobinopathy, etc.).
* Subjects with hemophilia or coagulation disorder, who are at increased risk of serious bleeding during intramuscular injection.
* Subjects who had an acute fever with body temperature > 38.0 ºC within 72 hours prior to administration of the study vaccine.
* Subjects who had received another vaccine within 28 days before administration of the study vaccine or are planning to receive another vaccine during the study.
* Subjects who had received immunosuppressants or immune modifying drugs within 3 months prior to the investigational product vaccination.

  1. Azathioprine, cyclosporin, interferon, G-CSF, tacrolimus, everolimus, sirolimus, etc.
  2. High dose corticosteroids (a subject taking high doses, which is defined as 2mg/kg/day or higher of prednisolone administered for longer than 14 consecutive days, is not eligible for this study. The use of inhaled, nasal and topical corticosteroids is allowed, regardless of doses).
* Subjects who had previously received immunoglobulin or blood-derived products within the last 3 months prior to administration of the study vaccine, or are scheduled to receive a treatment with blood-derived products during the study.
* Subjects who had participated in another clinical trial within the 30 days before administration of the study vaccine.
* Female subjects of childbearing potential who do not agree to use an acceptable method of birth control* for this study during the study period.

  * Medically acceptable methods of birth control: condom, injectable or implantable contraceptives, intrauterine device, or oral contraceptives, etc.
* Subjects with other clinically significant medical or psychiatric illness who in the investigator's opinion, are not be suitable for the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1794 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IL-YANG Quadrivalent Influenza Vaccine | IL-YANG Flu Vaccine Prefilled Syringe | IL-YANG Trivalent Influenza Vaccine
Started | 1197 | 298 | 299
Completed | 1186 | 296 | 296
Not Completed | 11 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IL-YANG Quadrivalent Influenza Vaccine | IL-YANG Flu Vaccine Prefilled Syringe | IL-YANG Trivalent Influenza Vaccine | Total
Number analyzed (Participants) | 1197 | 298 | 299 | 1794
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1015 | 254 | 253 | 1522
  >=65 years | 182 | 44 | 46 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (14.5) | 44.5 (14.7) | 45.7 (14.6) | 44.8 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 812 | 208 | 204 | 1224
  Male | 385 | 90 | 95 | 570

OUTCOME MEASURES:

1. Primary Outcome: Rate of Healthy Adults Aged ≥19 Years With Seroconversion
Description: Seroconversion is defined as follows. (Case 1) A pre-vaccination (Day 0) HI antibody titer < 1:10 and a post-vaccination (Day 28) HI antibody titer ≥ 1: 40. or (Case 2) a pre-vaccination (Day 0) HI antibody titer ≥ 1:10 and a minimum four-fold rise in post-vaccination (Day 28) HI antibody titer.
Time Frame: Day 28
Population: The immunogenicity data obtained from the study subjects were analyzed primarily in the Per Protocol Set that was consists of subjects who had at least one dose of the investigational product and from whom post-treatment primary efficacy endpoint data, and have completed the study up to Visit 3 without a major protocol violation.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | IL-YANG Quadrivalent Influenza Vaccine | IL-YANG Flu Vaccine Prefilled Syringe | IL-YANG Trivalent Influenza Vaccine
Number analyzed (Participants) | 1175 | 293 | 294
percentage of subjects
  A/H1N1 | 47.7 [44.9 to 50.6] | 49.5 [43.6 to 55.4] | 49.0 [43.1 to 54.8]
  A/H3N2 | 78.7 [76.3 to 81.0] | 81.6 [76.6 to 85.8] | 77.9 [72.7 to 82.5]
  B/Yamagata | 51.8 [48.9 to 54.7] | 54.9 [49.1 to 60.7] | 23.1 [18.4 to 28.4]
  B/Victoria | 47.7 [44.9 to 50.6] | 24.2 [19.4 to 29.6] | 54.8 [48.9 to 60.5]

2. Primary Outcome: Rate of Healthy Adults Aged ≥19 Years With Seroprotection
Description: Seroprotection: A post-vaccination (Day 28) HI antibody titer ≥ 1:40.
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | IL-YANG Quadrivalent Influenza Vaccine | IL-YANG Flu Vaccine Prefilled Syringe | IL-YANG Trivalent Influenza Vaccine
Number analyzed (Participants) | 1175 | 293 | 294
percentage of subjects
  A/H1N1 | 88.2 [86.2 to 90.0] | 89.4 [85.3 to 92.7] | 87.1 [82.7 to 90.7]
  A/H3N2 | 90.0 [88.1 to 91.6] | 92.5 [88.9 to 95.2] | 89.5 [85.4 to 92.7]
  B/Yamagata | 86.3 [84.2 to 88.2] | 88.4 [84.2 to 91.8] | 64.6 [58.9 to 70.1]
  B/Victoria | 84.9 [82.8 to 86.9] | 69.3 [63.7 to 74.5] | 85.7 [81.2 to 89.5]
Statistical Analysis 1: Comparison: IL-YANG Flu Vaccine Prefilled Syringe; To evaluate if the seroconversion (SCR) and seroprotection (SPR) rates on Day 28 after vaccination of IL-YANG Quadrivalent Influenza Vaccine Inj. meet the following criteria in all age groups of healthy male and female adults at the age of 19 or older; Test type: Equivalence — All statistical significance testing was performed at a two-sided significance level (α) of 5%. Exceptionally, non-inferiority was tested at a one-sided CI of 97.5%; p = 0.09135, ANCOVA

3. Secondary Outcome: Percentage of Subjects With SCR on Day 28 After Vaccination of the Investigational Product by Age Group
Description: The percentage of subjects with HI antibody SCR on Day 28 after vaccination of the investigational product was calculated and its 95% two-sided CI was presented for each strain by treatment group and by age group. The immunogenicity of the test vaccine was to be demonstrated if the lower limit of the 95% two-sided CI by age group was higher than the above mentioned criteria (40% for < 65 years of age, 30% for ≥ 65 years of age) in each treatment group.
Time Frame: Day 28
Population: Rate of healthy adults aged ≥19 ~ <65 years
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | IL-YANG Quadrivalent Influenza Vaccine | IL-YANG Flu Vaccine Prefilled Syringe | IL-YANG Trivalent Influenza Vaccine
Number analyzed (Participants) | 996 | 251 | 249
percentage of participants
  Strain H1N1 | 48.7 [45.5 to 51.8] | 51.8 [45.4 to 58.1] | 51.8 [45.4 to 58.2]
  Strain H3N2 | 80.3 [77.7 to 82.7] | 83.3 [78.1 to 87.7] | 78.7 [73.1 to 83.6]
  Strain B Yamagata | 52.3 [49.2 to 55.5] | 54.6 [48.2 to 60.9] | 24.5 [19.3 to 30.3]
  Strain B Victoria | 48.3 [45.1 to 51.4] | 27.5 [22.1 to 33.5] | 56.6 [50.2 to 62.9]

4. Secondary Outcome: Rate of Healthy Adults Aged ≥19 ~ <65 Years and ≥65 Years With Seroprotection, Respectively.
Description: Seroprotection is defined as follows. subjects who have a post-vaccination (Day 28) HI antibody titer ≥ 1: 40
Time Frame: Day 28
Population: Rate of healthy adults aged ≥65 years
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | IL-YANG Quadrivalent Influenza Vaccine | IL-YANG Flu Vaccine Prefilled Syringe | IL-YANG Trivalent Influenza Vaccine
Number analyzed (Participants) | 179 | 42 | 45
percentage of participants
  Strain H1N1 | 42.5 [35.1 to 50.1] | 35.7 [21.6 to 52.0] | 33.3 [20.0 to 49.0]
  Strain H3N2 | 69.8 [62.5 to 76.5] | 71.4 [55.4 to 84.3] | 73.3 [58.1 to 85.4]
  Strain B Yamagata | 49.2 [41.6 to 56.7] | 57.1 [41.0 to 72.3] | 15.6 [6.5 to 29.5]
  Strain B Victoria | 44.7 [37.3 to 52.3] | 4.8 [0.6 to 16.2] | 44.4 [29.6 to 60.0]

5. Secondary Outcome: Geometric Mean Titer as Measured by HI Antibody Titer on Day 28 After Vaccination of the Investigational Product (GMTcomparator/GMTtest Vaccine).
Time Frame: Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- IL-YANG Flu Vaccine Prefilled Syringe.IL-YANG Trivalent Influe: This TIV is included the B/Yamagata strain, and it was approved for commercial sale by MFDS.
  IL-YANG Flu Vaccine Prefilled Syringe: A single 0.5mL dose administrated as an intramuscular injection.
Arm/Group | IL-YANG Quadrivalent Influenza Vaccine | IL-YANG Flu Vaccine Prefilled Syringe.IL-YANG Trivalent Influe
Number analyzed (Participants) | 1175 | 587
Titer
  Strain H1N1 | 82.2 [77.8 to 86.9] | 85.1 [78.4 to 92.3]
  Strain H3N2 | 127.6 [119.5 to 136.2] | 130.6 [119.1 to 143.2]
  Strain B Yamagata | 74.3 [70.5 to 78.3] | 75.9 [67.9 to 85.0]
  Strain B Victoria | 60.1 [57.5 to 62.9] | 62.0 [56.5 to 68.1]

6. Secondary Outcome: Difference of Seroconversion Rate(SCR) of HI Antibody Titer After 28days Vaccination(SCRcomparator-SCRtest Vaccine)
Description: The IL-YANG Quadrivalent Influenza Vaccine contain two types of B strain, while two kinds of Trivalent Influenza Vaccine contain each type of B strain. Primary outcome was about seroconversion and seroprotection rate of HI antibody, so each results of 3 kinds of vaccine was described. Considering the cross-reaction between two types of B strain, the analysis was designed in a way that the SCR/SPR of the B strains can be compared, respectively.
  However, secondary outcome, unlike the primary outcome, is expressed as a ratio(difference of seroconversion rate). So, the above factors were not to be consider.
  All methods of analysis are comply with the request of MFDS, and the result data that may make you confuse will be delete.
Time Frame: Day 28
Population: Please see "Outcome Measure Description" and "Arm/Group Description"above.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- IL-YANG Trivalent Vaccine (Combined): This Arm/Group is combination of "IL-YANG Flu Vaccine Prefilled Syringe" and "IL-YANG Trivalent Influenza Vaccine" Arm/Group.
  -Reason that the two arms were combined IL-YANG Flu Vaccine Prefilled Syringe: contains H1N1, H3N2 and Yamagata strain. IL-YANG Trivalent Influenza Vaccine: includes H1N1, H3N2 and Victoria strain.
  -> To be used the above two trivalent vaccines as a control for the Quadrivalent vaccine, the results of seroconversion rate of above two trivalent vaccine was combined.
Arm/Group | IL-YANG Trivalent Vaccine (Combined) | IL-YANG Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 587 | 1175
percentage of participants
  Strain H1N1 | 49.2 [45.1 to 53.4] | 47.7 [44.9 to 50.6]
  Strain H3N2 | 79.7 [76.2 to 82.9] | 78.7 [76.3 to 81.0]
  Strain B Yamagata | 54.9 [49.1 to 60.7] | 51.8 [48.9 to 54.7]
  Strain B Victoria | 54.8 [48.9 to 60.5] | 47.7 [44.9 to 50.6]

7. Secondary Outcome: Geometric Mean Titer as Measured by HI Antibody Titer Before (Day 0) and on Day 28 After Vaccination of the Investigational Product.
Time Frame: Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | IL-YANG Quadrivalent Influenza Vaccine | IL-YANG Flu Vaccine Prefilled Syringe | IL-YANG Trivalent Influenza Vaccine
Number analyzed (Participants) | 1175 | 293 | 294
Titer
  Strain H1N1 | 82.2 [77.8 to 86.9] | 89.8 [79.7 to 101.3] | 80.6 [72.1 to 90.0]
  Strain H3N2 | 127.6 [119.5 to 136.2] | 135.6 [118.7 to 154.9] | 125.8 [110.7 to 143.0]
  Strain B Yamagata | 74.3 [70.5 to 78.3] | 75.9 [67.9 to 85.0] | 44.0 [39.6 to 48.7]
  Strain B Victoria | 60.1 [57.5 to 62.9] | 41.2 [37.6 to 45.2] | 62.0 [56.5 to 68.1]

8. Secondary Outcome: Geometric Mean Ratio as Measured by HI Antibody Titer Before (Day 0) and on Day 28 After Vaccination of the Investigational Product.
Time Frame: Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of GMT titer
Arm/Group | IL-YANG Quadrivalent Influenza Vaccine | IL-YANG Flu Vaccine Prefilled Syringe | IL-YANG Trivalent Influenza Vaccine
Number analyzed (Participants) | 1175 | 293 | 294
Ratio of GMT titer
  Strain H1N1 | 3.9 [3.6 to 4.2] | 4.1 [3.5 to 4.8] | 3.7 [3.1 to 4.3]
  Strain H3N2 | 9.5 [8.8 to 10.2] | 10.9 [9.5 to 12.6] | 9.8 [8.5 to 11.4]
  Strain B Yamagata | 3.3 [3.1 to 3.5] | 3.5 [3.1 to 3.9] | 2.0 [1.8 to 2.2]
  Strain B Victoria | 2.9 [2.8 to 3.1] | 2.1 [1.9 to 2.2] | 3.0 [2.7 to 3.3]

ADVERSE EVENTS:
Description: Safety set consists of all randomized subjects who had at least one dose of the investigational product. A subject who was randomized in this study but was withdrawn prior to vaccination of the investigational product was excluded from the safety set. There was 3-subject withdrawn prior to vaccination from 1197 enrolled subjects.
Arm/Group | IL-YANG Quadrivalent Influenza Vaccine | IL-YANG Flu Vaccine Prefilled Syringe | IL-YANG Trivalent Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 0/1194 | 2/298 | 1/299
Other Adverse Events (participants affected / at risk) | 0/1194 | 0/298 | 0/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IL-YANG Quadrivalent Influenza Vaccine (N=1194) | IL-YANG Flu Vaccine Prefilled Syringe (N=298) | IL-YANG Trivalent Influenza Vaccine (N=299)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No